CLINICAL TRIAL: NCT01891981
Title: Phase I/II Study of Moxetumomab Pasudotox in Patients With Relapsed and/or Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study of Moxetumomab Pasudotox in Patients With Relapsed and/or Refractory Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Ph I Exempt as it did not proceed to the Phase II terminated early by the supporter
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1143; NCI-2013-02207 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Lymphoblastic Leukemia; ALL; Relapsed and/or refractory; Moxetumomab Pasudotox; Maximum tolerated dose; MTD
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moxetumomab Pasudotox (Experimental): Phase I Starting Dose: 30 µg/kg by vein every other day for 6 doses on Days 1, 3, 5, 7, 9, and 11 of each 21-day cycle.
  Phase II Starting Dose: Maximum tolerated dose from Phase I.
  Interventions: Drug: Moxetumomab Pasudotox

INTERVENTIONS:
Drug: Moxetumomab Pasudotox — Phase I Starting Dose: 30 µg/kg by vein every other day for 6 doses on Days 1, 3, 5, 7, 9, and 11 of each 21-day cycle.
  Phase II Starting Dose: Maximum tolerated dose from Phase I.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of moxetumomab pasudotox that can be given to patients with relapsed and/or refractory ALL.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of 3-6 participants will be enrolled in the Phase 1 portion of the study.

If you are in Phase 1, the dose of moxetumomab pasudotox you receive will depend on when you join the study. The first group will receive the lowest dose level of moxetumomab pasudotox. Each additional group will receive a higher dose than the previous group, if no intolerable side effects were seen.

If you are in Phase 2, you will receive the highest dose of moxetumomab pasudotox found to be safe in the Phase 1 portion of the study.

Study Drug Administration:

You will receive moxetumomab pasudotox by vein on Days 1, 3, 5, 7, 9, and 11 of each 21-day cycle. You may be treated in the hospital for the first cycle. If your doctor thinks it is needed, the length of study cycles may be changed.

You may receive drugs to control side effects one hour before your dose of the study drug and up to 12 hours after your dose of the study drug. You may also receive fluids for hydration before and after your dose of the study drug.

Study Visits:

Every week during Cycle 1, blood (about 1 tablespoon) will be drawn for routine tests.

Within 1 week before Day 1 of each study cycle:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have an eye exam.
* Blood (about 2 teaspoons) will be drawn to test for drug antibodies.

On Day 1 (1st dose) of Cycle 1, before and right after your first dose of study drug and then 4-5 more times over the next 8 hours, blood (about 1/2 teaspoons each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. At the 6th dose, blood (about 1/2 teaspoon each time) will be drawn before and right after your dose of study drug for PK testing. PK testing for the 1st and 6th dose will be repeated for Cycle 2 and every 4th treatment cycle until the end of treatment.

If the doctor thinks the disease is responding to the study drug, blood (about 1 tablespoon) will be drawn at least 1 time every week for routine tests.

Between Days 14-21 (+/- 7 days) of Cycle 1, you will have a bone marrow biopsy/aspiration. You will have additional bone marrow biopsy/aspirations every 2-4 cycles after that, and then every 3 months for up to 1 year during the follow-up period.

At the end of each cycle, urine will be collected for routine tests.

After your last dose of study drug, blood (about 2 teaspoons) will be drawn to test for drug antibodies.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. If your doctor thinks the disease is responding, you may receive up to 6 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-Up Visit:

About 30 days after the last dose of the study drug, you will be asked to return to the clinic for follow-up tests. During this visit, you may have blood drawn and other tests performed to check the status of the disease, to test for drug antibodies, and to check your health.

If you cannot come to MD Anderson, you will be contacted by phone and asked about your health.

This is an investigational study. Moxetumomab pasudotox is not FDA approved or commercially available. At this time, it is being used for research purposes only.

Up to 60 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years or older with previously treated ALL (relapsed and/or refractory after prior therapy); patients with relapsed/refractory biphenotypic leukemia expressing the appropriate antigen (CD22) are also eligible to participate, Pediatric patients younger than 18 may be considered with sponsor approval once the MTD has been established in the adult population.
2. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
3. Adequate liver function (bilirubin less than or equal to 1.5 mg/dL and serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) less than or equal 2.5 x upper limit of normal (ULN), unless considered due to tumor or hemolysis), and renal function ( Calculated CrCl of greater than or equal to 50 or serum creatinine less than 2 x ULN.) Even if organ function abnormalities are considered due to tumor, the upper limit for bilirubin is less than or equal to 2.0 mg/dL (unless due to hemolysis or Gilbert's disease, i.e. mainly indirect bilirubin) and creatinine less than or equal 2 mg/dL
4. Provision of written informed consent.

Exclusion Criteria:

1. Patient with active heart disease (NYHA class greater than or equal to 2 as assessed by history and physical examination).
2. Patients with a cardiac ejection fraction (as measured by either multigated radionuclide angiography (MUGA) or echocardiogram) less than 40%
3. Patients with active hepatitis
4. Pregnant or breast-feeding women. Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days of start of treatment.
5. prior radioimmunotherapy within 3 years of enrollment
6. serum albumin less than 2g/dL
7. oxygen saturation at rest by pulse oximetry less than 88% or PaO2 less than or equal to 55mm Hg
8. history of microangiopathic hemolysis, TTP or HUS.
9. symptomatic central nervous system (CNS) involvement
10. Less than 100 days post -transplant or any evidence of active graft-versus-host disease (GVHD)
11. systemic chemotherapy less than 14 days prior; however treatment may start earlier if there is evidence of rapidly progressive disease if approved by the Principal Investigator
12. monoclonal antibody therapy less than 1 month
13. investigational agents within 28 days of dosing; however treatment may start earlier if there is evidence of rapidly progressive disease if approved by the Principal Investigator
14. HIV+/AIDS
15. history of exposure to pseudomonas exotoxin containing molecule
16. Patients with active lung infection or active pulmonary edema.
17. Patients with laboratory findings consistent with Grade equal to greater than 3 disseminated intravascular coagulation (DIC) or any Grade 2 DIC that does not correct.
18. Patients with clinically significant ophthalmologic findings (as determined by an ophthalmologist) during screening should be excluded from the trial
19. Pre-treatment greater than corrected QT interval (QTc) interval of 490 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Moxetumomab | After second 21 day cycle
  Maximum tolerated dose defined as the highest dose level in which 6 patients have been evaluated for toxicity and fewer than 2 dose limiting toxicities (DLTs) were observed. A non-hematologic DLT defined as a clinically significant Grade 3 or 4 adverse event or abnormal laboratory value assessed by treating physician as related to study drug (and unrelated to disease progression, intercurrent illness, or concomitant medications) occurring during the first 21(+/- 2) days on study. A hematologic dose-limiting toxicity defined as severe myelosuppression with a hypoplastic marrow with less than 5% cellularity and no evidence of leukemia 42 days from start of therapy.

SECONDARY OUTCOMES:
Overall Response Rate | After second 21 day cycle
  Primary efficacy outcome is overall response rate (including CR, CRi and PR). Complete remission (CR): Neutrophil count > 1.0 x109/L, platelet count >100x109/L, and normal marrow differential (< 5% blasts). Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recovery of counts (platelets < 100 x 109/L; neutrophils < 1 x 109/L). Partial remission (PR): Peripheral blood count recovery as for CR, but with decrease in marrow blasts of > 50% and not more than 25% abnormal cells in the marrow. Kaplan and Meier product limit method used to estimate the event-free survival (EFS) and overall survival (OS) and a 95% confidence interval for the median EFS and OS provided. Univariate and multivariate Cox proportional hazards regression model used to identify prognostic factors for EFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Muller F, Cunningham T, Stookey S, Tai CH, Burkett S, Jailwala P, Stetler Stevenson M, Cam MC, Wayne AS, Pastan I. 5-Azacytidine prevents relapse and produces long-term complete remissions in leukemia xenografts treated with Moxetumomab pasudotox. Proc Natl Acad Sci U S A. 2018 Feb 20;115(8):E1867-E1875. doi: 10.1073/pnas.1714512115. Epub 2018 Feb 5. PMID 29432154
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org